CLINICAL TRIAL: NCT04289987
Title: A Randomized, Double-blinded, Placebo-controlled, Parallel, Multicenter, Phase 2b Study to Evaluate the Efficacy and Safety of CVI-HBV-002 in Patients With Chronic Hepatitis B Taking Tenofovir
Brief Title: A Study to Evaluate the Efficacy and Safety of Therapeutic Hepatitis B Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHA Vaccine Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVI-HBV-002-CT1901
Record Dates: First submitted 2020-02-22; First posted 2020-02-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CVI-HBV-002 (Experimental): * CVI-HBV-002 1.0mL(20ug/dose)
  * Intramuscular injection at Baseline, Week 2, 4, 8, 12, 16, 20 / total 7 doses
  Interventions: Biological: CVI-HBV-002
- Normal Saline (Placebo Comparator): * Normal Saline Choonwae Inj. 1.0 mL
  * Intramuscular injection at Baseline, Week 2, 4, 8, 12, 16, 20 / total 7 doses
  Interventions: Biological: Normal Saline(placebo)

INTERVENTIONS:
Biological: CVI-HBV-002 — Investigational Product
  Arms: CVI-HBV-002
Biological: Normal Saline(placebo) — Investigational Product
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the investigational medicinal product CVI-HBV-002.

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo-controlled, parallel, multicenter, phase 2b study to evaluate the efficacy and safety of CVI-HBV-002 in patients with chronic hepatitis B taking Tenofovir disoproxil fumarate/Tenofovir disoproxil

ELIGIBILITY:
Inclusion Criteria:

1. Adult between 19 to 60 years of age
2. Those who have been diagnosed as chronic hepatitis B patients (e.g.HBsAg positive detected for 6 months or more)
3. Started treatment with Tenofovir Disoproxil Fumarate(TDF) or Tenofovir Diproxil(TD), oral HBV antiviral agent, for 6 months to 5 years.
4. HBsAg ≥ 100 IU/mL, HBV DNA ≤ 100 IU/mL at screening
5. HBV DNA ≤ 2000 IU/mL at screening
6. ALT ≤ Upper Limit of Normal) x 2 at screening
7. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures

Exclusion Criteria:

1. Patients with other hepatic disease other than chronic hepatitis B(e.g., hemochromatosis, Wilson disease, alcoholic liver disease, nonalcoholic steatohepatitis, alpha-1 antitrypsin deficiency, etc)
2. If any of the following laboratory tests were found at screening

   * Total bilirubin > Upper Limit of Normal x 2
   * Prothrombin time delayed more than 3 seconds than normal
   * Serum Albumin < 30 g/L (3 g/dL)
   * Hemoglobin < 9.0 g/dL eGFR < 60 mL/min (Cockcroft-Gault)
   * Absolute neutrophil count (ANC) < 1.5 x 10^9 /L (1500 /mm3)
   * Platelet count < 100 x 10^9 /L (100 x 10^3 /mm3)
   * Serum creatinine > 1.5 mg/dL
   * Serum amylase > 2 x ULN and Lipase > 2 x ULN
3. A history of ascites, jaundice, varicoses vein bleeding, hepatic encephalopathy, or other signs of liver failure
4. Treated with oral antiviral agents or interferon therapy other than TDF(or TD)
5. In case of receiving nephroxic drugs(Aminoglycosides, Amphotericin B, NSAIDs, etc.) within 14 days prior to screening
6. When hepatotoxic drugs(Erythromycin, Ketoconazole, Rifampin, Fluconazole, Dapsone, etc.) are administered within 14 days prior to screening
7. Patients with active bacterial, viral or fungal infections requiring systemic treatment
8. Patients diagnosed with Alpha-fetoprotein (AFP) >50 ng/mL or with Hepatocellular Carcinoma (HCC) in screening
9. Of those who have received immunosuppressive drugs within 6 months prior to screening, patients suspected of having decreased immunity by the judgment of the Investigator
10. Patients who have received high dose (prednisone 20mg or more*) systemic corticosteroids for a long period of time(consecutive 14 days or longer) within 3 months before screening (at the discretion of the investigator in case of local corticosteroids)

    * Corresponding to 125 mg of cortisone, 100 mg of hydrocortisone, 20 mg of prednisone, 16 mg of methylpreprednisolone, 16 mg of triamsynolone, 3 mg of dexamethasone and 2.4 mg of betametasone.
11. Patients who have been diagnosed with malignant tumors within 5 years before screening, or who have recurred malignant tumors(in case of benign tumors, if the Investigator considers that the progress of the clinical trial is not affected during the clinical trial)
12. Organ transplantation recipients
13. Patients with serious illnesses, such as heart failure, renal failure, and pancreatitis, other than liver disease
14. Patients with a history of serious heart disease (NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring treatment or unstable angina)
15. Patients with seizure disorders who require anticonvulsant therapy
16. HbA1c>7.5%
17. SBP≥140mmHg or DBP≥90mmHg
18. Patients infected with hepatitis C(HCV), hepatitis D(HDV) or human immunodeficiency virus(HIV)
19. A hypersensitivity or anaphylactic reaction to the components of the clinical trial drug or HBV vaccine components
20. Continued drinking(>21 units/week, 1 unit = 10g of pure alcohol) or alcohol dependence
21. Pregnancy or breastfeeding, or cannot agree with the approved method of contraception of the patient and partner during the clinical trial(e.g., infertility surgery, intrauterine contraceptive, oral contraceptive and concomitant use of diaphragm or condom, other hormonal delivery systems and concomitant use of diaphragm or condom)
22. Patients who are concerned about the deterioration of daily function due to mental illness or who cannot understand the purpose and method of this trial
23. Patient who has potential to severe febrile or systemic reaction
24. Patients who are scheduled to participate in other clinical trials after enrolling in this trial, or have participated in other clinical trials within 3 month of enrollment in this trial
25. Others those who are considered to be difficult to perform the clinical trial by the judgment of the Investigator

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of Mean Change in HBsAg(log10 IU/mL) | at week 48 from baseline
  To evaluate mean changes in serum HBsAg(log 10 IU/mL) for patients treated with CVI-HBV-002 or Placebo at Week 48 versus Baseline

SECONDARY OUTCOMES:
Evaluation of Mean changes in serum HBsAg(log 10 IU/mL) | at week 24 from baseline
  To evaluate mean changes in serum HBsAg(log 10 IU/mL) for patients treated with CVI-HBV-002 or Placebo at Week 24 versus Baseline
Proportion assessment of Participants With HBsAg loss | at weeks 24 and 48
  To evaluate proportion of subjects with HBsAg loss for patients treated with CVI-HBV-002 or Placebo at Weeks 24 and 48
Proportion assessment of Participants With HBsAg seroconversion | at weeks 24 and 48
  To evaluate proportion of subjects with HBsAg seroconversion for patients treated with CVI-HBV-002 or Placebo at Weeks 24 and 48
Proportion assessment of Participants With HBeAg loss | at Weeks 24 and 48
  To evaluate proportion of subjects with HBeAg loss for HBeAg positive patients treated with CVI-HBV-002 or Placebo at Weeks 24 and 48
Proportion assessment of Participants With HBeAg seroconversion | at weeks 24 and 48
  To evaluate proportion of subjects with HBeAg seroconversion for HBeAg positive patients treated with CVI-HBV-002 or Placebo at Weeks 24 and 48
Evaluation of changes in HBV specific T cell immunity | at weeks 12 and 24 from baseline
  Immune Response Rate of HBV specific T cell at Weeks 12 and 24 versus Baseline
Proportion assessment of Participants With Virologic breakthrough | Baseline to week 48
  Proportion of subjects with experiencing virologic breakthrough
Incidence assessment of Treatment-Emergent Adverse Evnent | Baseline to Week 48
  Safety and tolerability assessment through incidence of Treatment-Emergent Adverse Evnent after treatment of Investigational Product

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyeok Lee, Principal Investigator — Samsung Medical Center
Locations (9):
- South Korea (9):
  - Chung-ang University Hospital, Seoul, Dongjak-gu
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Korea University Guro Hospital, Seoul, Guro-gu
  - CHA University Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Severance Hospital, Seoul, Sedaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu
  - Soon Chung Hyang University Hospital Seoul, Seoul, Yongsan-gu